CLINICAL TRIAL: NCT03157960
Title: The Effect of Acute Fructose Load in Patients With Chronic Kidney Disease and Patients With Type 2 Diabetes Compared to Healthy Subjects
Brief Title: Effect of Acute Fructose Load in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Neda Rajamand Ekberg, M.D.,Ph.D, Karolinska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2011/1183-31/2
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Diseases; Diabetes Mellitus, Type 2
Keywords: Fructose; Uric acid; Oxidised LDL; Interleukin 6
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — blueberry extract; Carbonated Beverages; Fructose

STUDY DESIGN:
Intervention Model Description: Interventional study. Participant will on sex different occasions receive drinks containing fructose (fructose drink, coca-cola or blueberry drink) with and without the addition of a high-fat meal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Blueberry drink (Experimental): Participant will receive a blueberry drink containing 18 g of fructose and 14 g of glucose.
  Interventions: Other: Blueberry drink
- Blueberry and pizza (Experimental): Participant will receive a blueberry drink and a slice of pizza (170 grams; 22 g protein, 20 g fat and 50 g carbohydrate; 425 kCal)
  Interventions: Other: Blueberry and pizza
- Soft beverage (Experimental): Participant will receive a Soft beverage (Coca-cola containing 17,5 g fructose and 17,5 g glucose)
  Interventions: Other: Soft beverage
- Soft beverage and pizza (Experimental): Participant will receive a Soft beverage and a slice of pizza (170 grams; 22 g protein, 20 g fat and 50 g carbohydrate; 425 kCal)
  Interventions: Other: Soft beverage and pizza
- Fructose (Experimental): Participant will receive a drink containing 35 g of fructose
  Interventions: Other: Fructose
- Fructose and pizza (Experimental): Participant will receive a drink containing 35 g of fructose and a slice of pizza (170 grams; 22 g protein, 20 g fat and 50 g carbohydrate; 425 kCal)
  Interventions: Other: Fructose and pizza

INTERVENTIONS:
Other: Blueberry drink — Participant receive blueberry drink
  Arms: Blueberry drink
Other: Blueberry and pizza — Participant receive blueberry drink and a slice of pizza
  Arms: Blueberry and pizza
Other: Soft beverage — Participant receive a soft beverage drink
  Arms: Soft beverage
Other: Soft beverage and pizza — Participant receive a soft beverage drink and a slice of pizza
  Arms: Soft beverage and pizza
Other: Fructose — Participant receive a drink containing fructose
  Arms: Fructose
Other: Fructose and pizza — Participant receive a fructose drink and a slice of pizza
  Arms: Fructose and pizza

SUMMARY:
The metabolism of the monosaccharide fructose is less controlled than the metabolism of glucose, which will result in the metabolic product uric acid. Elevated serum uric acid levels are associated with increased risk, or worsening, of chronic kidney disease. The mechanisms by which uric acid have detrimental effects are not well defined, but may include an increase in reactive oxygen species and subsequent inflammatory activity. The aim of this study is to investigate the effects of uric acid, markers of oxidative stress and markers of inflammation following a low fructose load reflecting normal conditions. This is an interventional study. On six different occasions patients with chronic kidney disease, patients with type 2 diabetes and healthy controls will receive Blueberry drink, Coca-Cola or pure Fructose drink with similar amount of carbohydrates (140 kcal) with and without a high fat meal represented by a pizza (425 kcal).Serum samples and urinary samples will be collected.

DETAILED DESCRIPTION:
Fructose is a monosaccharide present naturally in foods as fruit, vegetables and honey. In fruit, vegetables and table sugar it is also present as a disaccharide (sucrose), where it is joined with glucose. The intake of fructose has increased dramatically in the last decades. The increase is attributed to the use of free fructose as a sweetener at higher concentrations than naturally occurring in food, where beverages as soft-drinks seem to be the largest contributor to present consumption. Fructose has a low glycemic index and thus helps maintain glycemic control, a property that led to the belief that it was beneficial as a sweetener for those with diabetes.

The body's capacity of absorbing fructose is limited and varies depending on age, health and co-ingested foods. Glucose is the dietary factor that has largest impact on fructose absorption, but animal studies also indicate that saturated fat increase absorption. It has been observed that the maximum fructose absorbing capacity varies between 5 and 50 g when consumed as a single dose. Individuals with type 2 diabetes seems to have a larger capacity to absorb fructose and they have higher levels of fructose in serum and urine when compared to those without diabetes.

Fructose is absorbed in the small intestine by the fructose specific transporter GLUT5. It is further transported to the liver through the portal vein, where it is absorbed and metabolized by liver cells. The metabolism of fructose is independent of insulin. Although some fructose is metabolized by the enterocytes in the small intestine, the liver metabolize the majority of ingested fructose, in comparison to about 15-30% of ingested glucose. The metabolism of fructose differs from glucose in the sense that it is less controlled. While glucose metabolism is regulated by the energy status of the cell and portal glucose concentrations, fructose metabolism lacks control mechanisms leading to different metabolic products and effects.

In the metabolic pathway fructose can be oxidized, converted to glucose or lactic acid, or enter de novo lipogenesis. In the first hepatic metabolic step fructose is phosphorylated by fructokinase, a fructose specific enzyme with high activity, to fructose-1-phosphate. Fructokinase is not regulated by the energy status (ATP) of the cell, and fructose will therefore be metabolized in an unlimited way. This is in contrast to steps in the glycolysis where phosphofructokinase is regulated by ATP. Due to the rapid phosphorylation of fructose, levels of ATP will be depleted followed by an increase in uric acid. An increase in reactive oxygen species will follow the formation of uric acid which may lead to inflammation in the endothelium and inflammatory activity in adipocytes. Animal models show that uric acid may also act directly on tubular cells in the kidney where it causes inflammation. Serum uric acid levels are moreover positively associated with renin activity and hypertension. Further, as fructose is metabolized in a less controlled way than glucose, a larger proportion of fructose is available for de novo lipogenesis (DNL). This may be due to that the capacity of the mitochondria is exceeded and acetyl-Coenzyme A will enter DNL instead of the citric acid cycle. This metabolic effect of glucose is considered as "particularly harmful". Whether glucose is co-ingested with fructose or not may have an impact on the metabolic effects as there will be an effect of secreted insulin. Insulin decreases production of glucose from fructose and stimulates the de novo lipogenesis pathway.

The increase in fructose consumption correlates closely with the rise in obesity, metabolic syndrome and diabetes. Long term consumption of fructose has been shown to cause increased uric acid in the body. Elevated serum uric acid levels are associated with risk of chronic kidney disease both among healthy subject and among those with diabetes. Among those with type 2 diabetes it has also been associated with progression of already established nephropathy.

It is estimated that 7.3 % of the adult population in Sweden is affected by diabetes and that the majority, 85 -90 %, constitutes of type 2 diabetes (T2D). T2D is considered to be one of the most common chronic diseases and the prevalence is expected to rise, and with that an increasing health and economic burden. Worldwide patterns indicate a growing burden as well, particularly in developing countries. T2D is a disease with multifactorial etiology and with complications such as cardiovascular and renal disease, blindness and amputation. Not only does diabetes affect quality of life, it also leads to premature death as life expectancy is reduced with as much as 15 years.

Diabetic nephropathy (DN) has become the most common cause of end-stage renal disease and the earliest sign of DN is presence of microalbuminuria. Further development of macroalbuminuria and a decline in glomerular filtration rate may follow. Among type 2 diabetics in Sweden it was observed that 20% developed albuminuria over the course of 5 years, and 11% developed renal impairment glomerular filtration rate (eGFR of < 60 mL/min/1.73m2, MDRD formula). Studies indicate that increased oxidative stress through different pathways may play a central role in the development of DN, and chronic hyperglycemia is the primary cause. But there are also other factors that increase oxidative stress and have an impact on development of renal disease, as for example free fatty acids and inflammation. The oxidative stress may cause damage to the renal milieu, as dysfunction of the endothelial cells within glomeruli and tissue injury of the tubule.

Factors related to disease management, as glycemic-, blood pressure- and lipid-control are important in protecting the kidney. Further, smoking cessation, energy balance for a healthy bodyweight and a healthy eating pattern are of importance. In regards of dietary composition, hyperglycemia and dyslipidemia is determined by the amount and quality of ingested carbohydrates and dietary fats. It has been suggested that postprandial hyperglycemia and hypertriglyceridemia triggers oxidative stress and causes inflammation, metabolic alterations associated with endothelial dysfunction. A prospective cohort conducted in 10 European countries, including Sweden (Malmö and Umeå) showed a protective effect of intake of vegetables, fruit and legumes against all-cause and cardiovascular mortality among those with diabetes. Possible mechanism is hypothesized to be attributed to the antioxidative properties. The anti-antioxidant and anti-inflammatory capacities of fruit and vegetables are mentioned as possible mechanisms.

Current Swedish dietary recommendation for diabetic's state that different diets as the Mediterranean and low carbohydrate diet etc. may be beneficial, while the scientific evidence for extremely low carbohydrate diet is yet too weak. They further state that single foods as fruit lower all-cause mortality and vegetables lowers the risk of cardiovascular mortality. Fructose is not discussed in the Swedish dietary recommendations. The American Diabetes Associations dietary recommendations do, however, state that fructose-containing beverages should be avoided due to its impact on metabolic profile.

The scientific evidence for the significance of diet on microvascular complications as kidney disease is scarce and there is a lack of studies on the effect of fruit and vegetables on diabetic nephropathy. This was also stated by Swedish Council on Health Technology Assessment (SBU) in a report published in 2010. SBU further emphasized the lack of dietary studies applicable to conditions in Sweden. Thus, considering the burden of type 2 diabetes and its related complications, the need for proposed studies is substantiate.

The overall aim of this study is to investigate the acute postprandial responses in uric acid, markers of oxidative stress and marker of inflammation after low fructose load with and without a high fat meal among patients with chronic kidney disease (CKD) and patients with type 2 diabetes (T2DM) with and without CKD compared to healthy controls (HC).

Patients with type 2 diabetes, patients with chronic kidney disease (CKD) and GFR <30 ml/min or dialysis, patients with type 2 diabetes and CKD and control subjects (n= 30 in each group) will be included. Participant will on sex different occasions receive drinks containing fructose with and without the addition of a high-fat meal. After including 8 patients with CKD, 8 patients with T2DM and 8 controls, the preliminary results will be presented.

ELIGIBILITY:
Inclusion Criteria:

* GFR <30 ml/min or >3 months of dialysis for patients with CKD
* Patients with type 2 diabetes with and without CKD
* Controls without diabetes type 2 or CKD

Exclusion Criteria:

* HbA1c > 100 mmol/mol.
* Signs of fluid overload
* Inability to understand the information provided for the study.
* Ongoing inflammatory disease or infection,
* Treatment with allopurinol or other uric acid lowering agents a

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in uric acid (µmol/L) | 2 hours for only drink and 4 hours for drink and a high fat meal
  Change in uric acid after intervention compared to the levels Before the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stenvinkel, professor, Study Director — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kolderup A, Svihus B. Fructose Metabolism and Relation to Atherosclerosis, Type 2 Diabetes, and Obesity. J Nutr Metab. 2015;2015:823081. doi: 10.1155/2015/823081. Epub 2015 Jun 14. PMID 26199742
- [Background] Tappy L, Le KA. Metabolic effects of fructose and the worldwide increase in obesity. Physiol Rev. 2010 Jan;90(1):23-46. doi: 10.1152/physrev.00019.2009. PMID 20086073
- [Background] Dyer J, Wood IS, Palejwala A, Ellis A, Shirazi-Beechey SP. Expression of monosaccharide transporters in intestine of diabetic humans. Am J Physiol Gastrointest Liver Physiol. 2002 Feb;282(2):G241-8. doi: 10.1152/ajpgi.00310.2001. PMID 11804845
- [Background] Bjornstad P, Lanaspa MA, Ishimoto T, Kosugi T, Kume S, Jalal D, Maahs DM, Snell-Bergeon JK, Johnson RJ, Nakagawa T. Fructose and uric acid in diabetic nephropathy. Diabetologia. 2015 Sep;58(9):1993-2002. doi: 10.1007/s00125-015-3650-4. Epub 2015 Jun 7. PMID 26049401
- [Background] Mayes PA. Intermediary metabolism of fructose. Am J Clin Nutr. 1993 Nov;58(5 Suppl):754S-765S. doi: 10.1093/ajcn/58.5.754S. PMID 8213607
- [Background] Jia G, Aroor AR, Whaley-Connell AT, Sowers JR. Fructose and uric acid: is there a role in endothelial function? Curr Hypertens Rep. 2014 Jun;16(6):434. doi: 10.1007/s11906-014-0434-z. PMID 24760443
- [Background] Feig DI, Kang DH, Johnson RJ. Uric acid and cardiovascular risk. N Engl J Med. 2008 Oct 23;359(17):1811-21. doi: 10.1056/NEJMra0800885. No abstract available. PMID 18946066
- [Background] Hovind P, Rossing P, Johnson RJ, Parving HH. Serum uric acid as a new player in the development of diabetic nephropathy. J Ren Nutr. 2011 Jan;21(1):124-7. doi: 10.1053/j.jrn.2010.10.024. PMID 21195935
- [Background] Riegersperger M, Covic A, Goldsmith D. Allopurinol, uric acid, and oxidative stress in cardiorenal disease. Int Urol Nephrol. 2011 Jun;43(2):441-9. doi: 10.1007/s11255-011-9929-6. Epub 2011 Mar 10. PMID 21547469
- [Background] Soltani Z, Rasheed K, Kapusta DR, Reisin E. Potential role of uric acid in metabolic syndrome, hypertension, kidney injury, and cardiovascular diseases: is it time for reappraisal? Curr Hypertens Rep. 2013 Jun;15(3):175-81. doi: 10.1007/s11906-013-0344-5. PMID 23588856
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] Zhang P, Zhang X, Brown J, Vistisen D, Sicree R, Shaw J, Nichols G. Global healthcare expenditure on diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Mar;87(3):293-301. doi: 10.1016/j.diabres.2010.01.026. Epub 2010 Feb 19. PMID 20171754
- [Background] Davies MJ, Tringham JR, Troughton J, Khunti KK. Prevention of Type 2 diabetes mellitus. A review of the evidence and its application in a UK setting. Diabet Med. 2004 May;21(5):403-14. doi: 10.1111/j.1464-5491.2004.01176.x. PMID 15089783
- [Background] Singh DK, Winocour P, Farrington K. Oxidative stress in early diabetic nephropathy: fueling the fire. Nat Rev Endocrinol. 2011 Mar;7(3):176-84. doi: 10.1038/nrendo.2010.212. Epub 2010 Dec 14. PMID 21151200
- [Background] Shields J, Maxwell AP. Managing diabetic nephropathy. Clin Med (Lond). 2010 Oct;10(5):500-4. doi: 10.7861/clinmedicine.10-5-500. PMID 21117388
- [Background] Forbes JM, Cooper ME. Mechanisms of diabetic complications. Physiol Rev. 2013 Jan;93(1):137-88. doi: 10.1152/physrev.00045.2011. PMID 23303908
- [Background] Afghahi H, Cederholm J, Eliasson B, Zethelius B, Gudbjornsdottir S, Hadimeri H, Svensson MK. Risk factors for the development of albuminuria and renal impairment in type 2 diabetes--the Swedish National Diabetes Register (NDR). Nephrol Dial Transplant. 2011 Apr;26(4):1236-43. doi: 10.1093/ndt/gfq535. Epub 2010 Sep 3. PMID 20817668
- [Background] van Dijk C, Berl T. Pathogenesis of diabetic nephropathy. Rev Endocr Metab Disord. 2004 Aug;5(3):237-48. doi: 10.1023/B:REMD.0000032412.91984.ec. No abstract available. PMID 15211095
- [Background] Ahmad J. Management of diabetic nephropathy: Recent progress and future perspective. Diabetes Metab Syndr. 2015 Oct-Dec;9(4):343-58. doi: 10.1016/j.dsx.2015.02.008. Epub 2015 Mar 6. PMID 25845297
- [Background] Evert AB, Boucher JL, Cypress M, Dunbar SA, Franz MJ, Mayer-Davis EJ, Neumiller JJ, Nwankwo R, Verdi CL, Urbanski P, Yancy WS Jr. Nutrition therapy recommendations for the management of adults with diabetes. Diabetes Care. 2014 Jan;37 Suppl 1:S120-43. doi: 10.2337/dc14-S120. No abstract available. PMID 24357208
- [Background] O'Keefe JH, Gheewala NM, O'Keefe JO. Dietary strategies for improving post-prandial glucose, lipids, inflammation, and cardiovascular health. J Am Coll Cardiol. 2008 Jan 22;51(3):249-55. doi: 10.1016/j.jacc.2007.10.016. PMID 18206731